CLINICAL TRIAL: NCT06301503
Title: Postoperative Quality of Recovery After Combined Lumbar Plexus-Sciatic Nerve Block for Lower Extremity Orthopaedic Surgeries: A Double-Blind Randomised Controlled Trial
Brief Title: Postoperative Quality of Recovery After Combined Lumbar Plexus-Sciatic Nerve Block (LPB-SNB)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Udayana University (Other)
Responsible Party: Principal Investigator, Jeremia Alvian Wiranata, Anesthesiologist Resident, Udayana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0103/UN14.2.2.VII.14/LT/2024
Record Dates: First submitted 2024-03-02; First posted 2024-03-08 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Lower Extremity Surgery

STUDY DESIGN:
Intervention Model Description: One hundred participants are to be randomly assigned by a computer-generated random number table into two parallel groups and 1:1 allocation to either receive a combination of LPB-SNB or no block at all.
Who Masked: Participant, Outcomes Assessor
Masking Description: Numbers were prepared in sealed envelopes prepared by a third party not involved in the study to ensure allocation concealment, and handed over to the anesthetist performing the block before surgery. Both participants and outcome assessors would be blinded to the group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1. USG Guided Combined LPB-SNB with Isobaric Bupivacaine (Experimental): After completing the surgical procedure under spinal anaesthesia, participants are positioned in the lateral decubitus position with the side to be blocked facing upwards. Identification of the lumbar plexus nerves is carried out with ultrasound guidance using the trident approach. Under aseptic conditions, local anesthetic infiltration with 2% lidocaine (3ml)was given, and a lumbar plexus block (LPB) technique was performed by inserting a 100mm insulated nerve block needle through the transverse process, delivering a bolus of 0.25% isobaric bupivacaine (20ml).
  Without changing the participant's position, the sciatic nerve is identified by the gluteal approach. After local anesthetic infiltration with 2% lidocaine (3ml), sciatic nerve block (SNB) was performed by inserting a 100 mm insulated nerve block needle to the sciatic nerve, delivering a bolus of 0.25% isobaric bupivacaine (20ml).
  Aspiration is carried out before injecting anaesthetic agent on each puncture sites.
  Interventions: Drug: USG Guided Combined LPB-SNB with Isobaric Bupivacaine
- 2. Control (Active Comparator): Postoperatively, participants in this group was positioned in the lateral decubitus position and both the lumbar plexus and sciatic nerves were identified using ultrasound. Local anesthetic infiltration was given at both puncture sites, but participants of this group did not receive a combination of LPB-SNB with bupivacaine.
  Interventions: Drug: Control

INTERVENTIONS:
Drug: USG Guided Combined LPB-SNB with Isobaric Bupivacaine — Local anesthetic infiltration of 2% lidocaine (3ml) along with injection anaesthetic agent consisting of isobaric bupivacaine 0.25% (20 ml)
  Other Names: LPB; SNB; Lumbar Plexus Block; Sciatic Nerve Block; Psoas Compartment Block (PCB); PCB
  Arms: 1. USG Guided Combined LPB-SNB with Isobaric Bupivacaine
Drug: Control — Local anesthetic infiltration of 2% lidocaine (3ml)
  Other Names: PCA-Only; Non-Block
  Arms: 2. Control

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of lumbar plexus-sciatic nerve block (LPB-SNB) by comparing the postoperative quality of recovery as assessed by the Quality of Recovery-40 (QoR-40) questionnaire, in patients who received a combination of LPB-SNB versus patients who received the traditional intravenous opioid, after lower extremity orthopaedic surgeries with spinal anaesthesia.

The main questions it aims to answer are:

* Will there be a significant difference in QoR-40 scores between both groups?
* Will the combined LPB-SNB significantly reduces opioid consumption within the first 24 hours?
* Will the combined LPB-SNB significantly increases postoperative duration of analgesia?

Participants will:

* Receive a coded sealed opaque envelope containing their randomly allocated intervention group; first group receives a combination of lumbar plexus-sciatic nerve block, while the second group receives no block at all. This information would not be disclosed to the participants.
* Receive an explanation on how to use the patient controlled analgesia (PCA) to deliver intravenous opioid, and instructions on filling in the QoR-40 questionnaire.

Researchers will then compare the results between both groups to see if the combined lumbar plexus-sciatic nerve block successfully provides adequate analgesia and enhance postoperative quality of recovery after lower extremity orthopaedic surgeries.

DETAILED DESCRIPTION:
Following lower extremity orthopaedic surgeries, acute postoperative pain management plays a crucial on each patient's quality of recovery. Postoperative pain are usually classified as nociceptive, neuropathic, mixed, psychogenic, or idiopathic and so, a single treatment might be insufficient to treat it adequately. Multimodal analgesia, encompassing techniques such as the neuraxial blockade, peripheral nerve blocks, infiltration, patient-controlled opioid analgesia, and nonsteroidal anti-inflammatory drugs (NSAIDS), has been extensively investigated with aims to relieve postoperative pain.

Lumbar Plexus Block (LPB) and Sciatic Nerve Block (SNB) are peripheral nerve block techniques consisting of the two large nerve branches that innervate the lower leg area. The combination of these two blocks (LPB-SNB), guided by ultrasonography (USG), blocks pain sensation throughout the lower extremity, and has been studied as an effective multimodal analgesia technique to relieve postoperative pain. This technique can minimize postoperative pain and also reduce the amount of opioid consumption, thereby reducing the incidence of postoperative nausea and vomiting (PONV).

Patients' opinions of their medical care are the subject of an expanding array of assessment instruments being developed to gauge the level of postoperative recovery. The QoR-40 questionnaire is gaining popularity due to considerable validation of its utility in measuring quality of recovery. This questionnaire is appropriate for its intended use, responsive to changes in the therapeutic setting, and can yield reliable findings. The QoR-40 is a useful tool for assessing the anaesthesia and postoperative recovery quality in patients undergoing peripheral nerve blocks as well as in ordinary clinical practice. Nonetheless, there is currently limited research using the QoR-40 questionnaire to assess the quality of recovery in studies evaluating the efficacy of peripheral nerve blocks.

This randomised controlled, double-blind and single-center trial will be conducted in a tertiary care hospital with aims of evaluating the efficacy of combined LPB-SNB compared to the traditional intravenous opioid in providing adequate analgesia after lower extremity orthopaedic surgeries with spinal anaesthesia with its primary outcome being the patient's postoperative quality of recovery as assessed by the QoR-40 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing lower extremity orthopaedic surgery with spinal anaesthesia
* Patients aged between 18-65 years
* Patients with American Society of Anesthesiologists (ASA) physical status classification of I-III
* Patients with a body mass index (BMI) between 18-30 kg/m2

Exclusion Criteria:

* Patients with a history of allergy towards the local anaesthetic agents used
* Patients with contraindication to regional anaesthesia based on the American Society for Regional Anesthesia guidelines
* Patients with pre-existing mental or psychological disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-03-09 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Postoperative Quality of Recovery as assessed by the QoR-40 questionnaire | 24 hours postoperatively
  The QoR-40 questionnaire is gaining popularity due to considerable validation of its utility in measuring quality of recovery. The QoR-40 questionnaire has 40 questions divided into 5 assessment dimensions, namely comfort (12 questions), emotions (9 questions), physical independence (5 questions), support (8 questions) and pain (6 questions), where each question has a value of 1 to 5 based on the Likert scale.

SECONDARY OUTCOMES:
Postoperative Intravenous Opioid Consumption | 24 hours postoperatively
  Total opioid consumption within 24 hours after lower extremity orthopaedic surgery (in milligrams).
Postoperative Analgesia Duration | Within 24 hours postoperatively
  The duration of the postoperative analgesia, measured from the time the surgery was done (control group) or combined block was given (combined LPB-SNB group) till the time when participant first presses the PCA button in request of intravenous opioid (in minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremia A Wiranata, MD, Principal Investigator — Udayana University
Locations (1):
- Prof. Dr. I.G.N.G. Ngoerah General Hospital, Denpasar, Bali, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning from 6 months and ending in 2 years after online article publication
Access Criteria: Researchers who provide a methodologically sound proposal of related studies. Proposals should be directed to jeremiaalvian@student.unud.ac.id.
  To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Background] Touray ST, de Leeuw MA, Zuurmond WW, Perez RS. Psoas compartment block for lower extremity surgery: a meta-analysis. Br J Anaesth. 2008 Dec;101(6):750-60. doi: 10.1093/bja/aen298. Epub 2008 Oct 22. PMID 18945717
- [Background] Strid JMC, Sauter AR, Ullensvang K, Andersen MN, Daugaard M, Bendtsen MAF, Soballe K, Pedersen EM, Borglum J, Bendtsen TF. Ultrasound-guided lumbar plexus block in volunteers; a randomized controlled trial. Br J Anaesth. 2017 Mar 1;118(3):430-438. doi: 10.1093/bja/aew464. PMID 28203808
- [Result] Horasanli E, Gamli M, Pala Y, Erol M, Sahin F, Dikmen B. A comparison of epidural anesthesia and lumbar plexus-sciatic nerve blocks for knee surgery. Clinics (Sao Paulo). 2010;65(1):29-34. doi: 10.1590/S1807-59322010000100006. PMID 20126343
- [Result] Aissa I, Wartiti LE, Bouhaba N, Khallikane S, Moutaoukil M, Kartite N, Elkoundi A, Benakrout A, Chlouchi A, Elbouti A, Najout H, Grine A, Touab R, Zaizi A, Youssef J, Bakkali H, Balkhi H, Bensghir M. [Combined lumbar plexus-sciatic nerve block in the emergency surgery for pertrochanteric fracture: an alternative technique in patients at high risk of anaesthetic complications]. Pan Afr Med J. 2020 Sep 3;37:12. doi: 10.11604/pamj.2020.37.12.21392. eCollection 2020. French. PMID 33062115